CLINICAL TRIAL: NCT02803385
Title: Comparison of Efficacy of Patient Controlled Epidural Analgesia Versus Continuous Epidural Infusion Following Thoraco-abdominal Surgeries in Cancer Patients
Brief Title: Comparison of Patient Controlled & Continuous Epidural Analgesia in Thoraco-abdominal Surgeries in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, parmanand jain, Professor, Tata Memorial Centre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1681
Record Dates: First submitted 2016-06-08; First posted 2016-06-17 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Pain
Keywords: Patient Controlled Epidural Analgesia; Continous Epidural Infusion Analgesia
MeSH Terms: conditions — Pain | interventions — Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continous Epidural Analgesia (Active Comparator): Continuous epidural infusion at rate of 5-8 ml /hr based on maximum allowable safe dose as per body weight. The Patient Controlled Analgesia pump settings will be set at 0.1 ml per bolus with lockout interval of 20 minutes
  Interventions: Other: Continous Epidural Analgesia
- Patient Controlled Epidural Analgesia (Active Comparator): Patient controlled epidural analgesia in form of PCA pumps with continuous rate of 5-8ml/hour & demand dose of 2-3 ml p.r.n with a lock out interval of 20 minutes based on maximum allowable safe dose as per body weight .
  Interventions: Other: Patient Controlled Epidural Analgesia

INTERVENTIONS:
Other: Continous Epidural Analgesia — continuous epidural infusion at rate of 5-8 ml /hr based on maximum allowable safe dose as per body weight. The pump settings will be set at 0.1 ml per bolus with lockout interval of 20 minutes. Cross over to other group will occur after 36hours.
  Other Names: continous epidural infusion of local anesthetic with opioid
  Arms: Continous Epidural Analgesia
Other: Patient Controlled Epidural Analgesia — patient controlled epidural analgesia in form of Patient Controlled Analgesia pumps with continuous rate of 5-8ml/hour & demand dose of 2-3 ml p.r.n with a lock out interval of 20 minutes based on maximum allowable safe dose as per body weight .The group will have a cross over at 36 hours postop.
  Other Names: patient controlled boluses of local anesthetic with opioid
  Arms: Patient Controlled Epidural Analgesia

SUMMARY:
This study aims to compare the efficacy of pain control, the consumption of local anesthetic and opioids, side effects, and patient satisfaction between continuous epidural infusion and patient controlled epidural analgesia after thoraco-abdominal surgeries in cancer patients.

DETAILED DESCRIPTION:
Aim-

1. To compare the pain scores during rest and movement with continuous epidural infusion (CEI) vs. patient controlled epidural analgesia (PCEA)
2. To compare the incidence of side effects between 2 groups
3. Comparison of local anaesthetic and opioids requirement by PCA attempts and also rescue analgesia requirement.
4. To compare patient satisfaction with the two different modalities of pain management

Sample size- Based on our hospital data for postoperative pain management after thoraco-abdominal surgeries, it was found that 69.7 % patients experience moderate to severe pain (pain score 4-10) on first day postoperatively.

Considering a 50% reduction as meaningful, group sample size of 62 with 31 in each group was calculated using a chi square test. Assuming a 10% loss to follow up or drop outs from study we require 35 in each group with total sample size of 70.

Variables- age, sex, demographic factors, surgery, duration of surgery, pain score, nausea score, hypotension episode, pruritis, Vomiting episode, patients satisfaction score, requirement of rescue analgesia.

Analysis of variables:

Descriptive statistics will be used for data representation. The χ2 and Fisher's exact probability tests will be used to analyze the differences between qualitative data. Comparisons of two groups will be analyzed using the Independent sample t test or Mann-Whitney U test as per the distribution of data. A P-value less than 0.05 will be considered statistically significant. Patient satisfaction using verbal rating scale will be analysed using Mann-Whitney U test.

Methodology- Patient meeting inclusion criteria, 4 hours after surgery will be reassessed in absence of any post-operative exclusion criteria, patient will be randomized into either group as per a computer generated chart and study will start from this time.

Postoperative group A will receive continuous epidural infusion at rate of 5-8 ml /hr based on maximum allowable safe dose as per body weight[10]. The Patient Controlled Analgesia settings will be set at 0.1 ml per bolus with lockout interval of 20 minutes.

Group B will receive patient controlled epidural analgesia in form of Patient Controlled analgesia pumps with continuous rate of 5-8ml/hour & demand dose of 2-3 ml p.r.n with a lock out interval of 20 minutes based on maximum allowable safe dose as per body weight . Both the groups will have a cross over at 36 hours postop.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients, American Society of Anaesthesia class I-II, posted for thoraco-abdominal surgeries and planned for epidural catheter insertion for perioperative pain management, will be included. The surgeries will include gastrectomy, radical & revision cholecystectomy, whipples procedure, pancreatectomy, lobectomy, metastectomy, pneumonectomy will be included.

Exclusion Criteria:

1. Patients with contraindication to epidural catheter placement or use of opioids or local anesthetic
2. Patients with contraindication to use of rescue analgesia like paracetamol and diclofenac both in postoperative period
3. Multiple incision not covered with epidural like TTE, THE
4. Patients with failed epidural insertion
5. Patients with epidural band not covering the incision sites completely
6. Patient with hemodynamic instability leading to inability to use epidural within the first 4-6 hours.
7. Patient shifted on ventilator or needing ventilator support the within first 6-12 hours.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
To compare the pain scores during rest and movement with continuous epidural infusion (CEI) vs. patient controlled epidural analgesia (PCEA) | 72 hours
  pain scores to be assessed using Numerical Rating scale(1-10)

SECONDARY OUTCOMES:
To compare patient satisfaction between the two groups using Verbal Rating scale | 36 hours and 72 hours
To assess the incidence of side effects in both groups including hypotension, motor weakness, pruritus, nausea, vomiting and any other | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Parmanand Jain, MD, MNAMS, Principal Investigator — Professor; Sumitra Bakshi, MD, Study Chair — Professor; Ankita Lapalikar, MBBS, Study Chair — Student
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu SS, Allen HW, Olsson GL. Patient-controlled epidural analgesia with bupivacaine and fentanyl on hospital wards: prospective experience with 1,030 surgical patients. Anesthesiology. 1998 Mar;88(3):688-95. doi: 10.1097/00000542-199803000-00020. PMID 9523813
- [Result] Komatsu H, Matsumoto S, Mitsuhata H, Abe K, Toriyabe S. Comparison of patient-controlled epidural analgesia with and without background infusion after gastrectomy. Anesth Analg. 1998 Oct;87(4):907-10. doi: 10.1097/00000539-199810000-00030. PMID 9768792
- [Result] Standl T, Burmeister MA, Ohnesorge H, Wilhelm S, Striepke M, Gottschalk A, Horn EP, Schulte Am Esch J. Patient-controlled epidural analgesia reduces analgesic requirements compared to continuous epidural infusion after major abdominal surgery. Can J Anaesth. 2003 Mar;50(3):258-64. doi: 10.1007/BF03017795. PMID 12620949